CLINICAL TRIAL: NCT02307331
Title: RCT of the Sirius Stem Used in Conjunction With the Exceed ABT Cemented Cup and OptiPac/OptiVac Cement - Model Based RSA, Clinical and Radiographic Outcomes
Brief Title: RSA Study of Sirius Stem and Exceed Cup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sirius RSA study_JT
Record Dates: First submitted 2014-11-25; First posted 2014-12-04 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis
Keywords: Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Optivac and E1 (Other): Sirius stem used with Optivac mixed cement - Exceed Cup - E1 PE
  Interventions: Device: Optivac; Device: E1 (Exceed cup); Device: Sirius stem
- Optivac and Arcom (Other): Sirius stem used with Optivac mixed cement - Exceed Cup - Arcom PE
  Interventions: Device: Optivac; Device: Arcom (Exceed cup); Device: Sirius stem
- Optipac and E1 (Other): Sirius stem used with Optipac mixed cement - Exceed Cup - E1 PE
  Interventions: Device: Optipac; Device: E1 (Exceed cup)
- Optipac and Arcom (Other): Sirius stem used with Optipac mixed cement - Exceed Cup - Arcom PE
  Interventions: Device: Optipac; Device: Arcom (Exceed cup); Device: Sirius stem

INTERVENTIONS:
Device: Optivac — A vacuum mixing system for cement with mixing and collection under vacuum but open initial mixture of powder and monomer. Has been used since 1993 with excellent results
  Arms: Optivac and Arcom; Optivac and E1
Device: Optipac — A vacuum mixing system for cement with mixing and collection under vacuum but with a pre-packed mixing system allowing for an all closed system minimizing exposure for monomer fumes. This is a relatively new mixing system
  Arms: Optipac and Arcom; Optipac and E1
Device: Arcom (Exceed cup) — The Exceed cup is available in two type of advanced bearing polyethylene material: The first is the 'classic', long term proven ArCom, a conventional polyethylene
  Arms: Optipac and Arcom; Optivac and Arcom
Device: E1 (Exceed cup) — The Exceed cup is available in two type of advanced bearing polyethylene material: The new is a highly cross linked polyethylene with infusion of vitamin E1 to remove free radicals in order to reduce wear.
  Arms: Optipac and E1; Optivac and E1
Device: Sirius stem — A polished tapered stem
  Arms: Optipac and Arcom; Optivac and Arcom; Optivac and E1

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the Sirius Cemented Stem used in conjunction with the Exceed ABT Cemented Acetabular Cup, either with E1 or Arcom polyethylene, and OptiPac/OptiVac bone cement mixing systems.

DETAILED DESCRIPTION:
This is a comparative, prospective randomized Radiostereometry (RSA) study, lead on 48 patients in a single site.

All 48 patients will be pooled in a single group for the evaluation of the primary criterion for evaluation, but randomized into four groups for the evaluation of the secondary criteria for evaluation

The objectives of the study are to:

1. Demonstrate a comparable migration pattern as is described in published literature on other double tapered polished cemented stems
2. Measure wear pattern in the cup made of vitamin-E doped polyethylene or conventional Arcom polyethylene

2)Demonstrate non-inferiority of Optipac vs. Optivac cement mixing systems on the stem side 3)Evaluate the clinical outcome and survivorship of the implant

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are eligible for cemented total hip arthroplasty
2. Patients diagnosed with primary Osteoarthritis
3. Patients who are fit for elective surgery (ASA I - III)
4. Patients with a BMI between 16 and 40
5. Patients who are skeletally mature
6. Patients aged over 18 at the time of surgery
7. Patients willing to return for follow-up evaluations
8. Patients who have the ability to follow instructions
9. Patients with sufficient bone stock and quality

Exclusion Criteria:

1. Female patients who are pregnant or planning pregnancy during the course of the study (no use of adequate birth control)
2. Patients with diagnosed active infection
3. Patients with marked bone loss which could preclude or compromise adequate fixation of the device
4. Patients with Parkinson disease
5. Patients using immunosuppressive drugs
6. Patients with an immunosuppressive disease
7. Patients with BMI <16
8. Patient with BMI >40
9. Patients who are unfit for surgery (ASA IV - V)
10. Patients with acetabular or femoral osteotomy
11. Patients who had a THA on the contralateral side within last 6 months
12. Patients belonging to the vulnerable population: children, patients with mental

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Radiostereometry (RSA) - change in migration and wear over time | First postoperative day, 3 months, 1 year, 2 years and 5 years
  Prosthesis migration and cup wear are measured over time, from baseline directly postop up to 5years. Measures are given in change in mm (translation) and degrees (rotation) around x, y and z-axis.

SECONDARY OUTCOMES:
Conventional Radiography (Signs of radiolucent lines or obvious change of position will be measured in mm) | First postoperative day, 2 years and 5 years
  Signs of radiolucent lines or obvious change of position will be measured in mm
HOOS (Hip specific health questionnaire) | Preoperatively, 1 year, 2 years and 5 years
  Hip specific health questionnaire - HOOS
EQ5D | Preoperatively, 1 year, 2 years and 5 years
  General health questionnaire - EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Flivik, Md PhD, Principal Investigator — Dept of Orthopedics, Skane University Hospital, Lund University
Locations (1):
- Deot of Orthopedics, Skane University Hospital, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No